CLINICAL TRIAL: NCT06944483
Title: Same-day Radioembolization for Large HCC (>5cm) With Y90 Resin Microspheres : Multicenter Prospective Registry Study
Brief Title: Same-day Radioembolization for Large HCC
Acronym: ISTAR-01
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Cheol Kim, Clinical Professor, Seoul National University Hospital
Other Study IDs: 2503-051-1620
Record Dates: First submitted 2025-04-08; First posted 2025-04-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- same-day group: planning angiography, MAA scan, and radioembolization was performed in a single day
  Interventions: Procedure: same-day radioembolization

INTERVENTIONS:
Procedure: same-day radioembolization — On the day of the procedure, angiography is performed, followed by cone-beam CT of the hepatic artery. After injecting 99mTc-MAA into the hepatic artery, the patient is transferred to the nuclear medicine department for a lung shunt scan and lung SPECT/CT. The lung shunt fraction is determined using the planar images.
  Using diagnostic CT/MRI and 99mTc-MAA images, the treatment dose is calculated with the multi-compartment MIRD method. The acceptable range for tumor absorbed dose is ≥100 Gy, and the lung dose must be ≤15 Gy. The tumor absorbed dose must be at least 100 Gy and should ideally be within the range of 300 to 600 Gy. There is no upper limit for the tumor absorbed dose.

SUMMARY:
In patients who has no sign suggesting high lung shunt fraction (TIPS, hepatic vein invasion, hepatic vein enhancement on arterial phase, dysmorphic intratumoral vessel), planning angiography, MAA scan, and radioembolization are performed in a single day with SIR-Spheres. This prospective registry will prove that the selection criteria is accurate and same-day radioembolization is feasible and safe.

DETAILED DESCRIPTION:
SIR-Spheres (SIRTEX): A mother vial containing ≥7 GBq is delivered to the hospital, and the treatment team divides it into daughter vials with specific radiation activities tailored to the target vessels. This allows for same-day TARE, in which lung shunt evaluation, vessel identification, dose calculation, and microsphere injection are all conducted on the same day.

This approach is referred to as same-day TARE.

To implement same-day TARE effectively, it is crucial to carefully select patients who are expected to have a low lung shunt fraction. This helps minimize the waste of pre-ordered SIR-Spheres vials that would otherwise go unused. Factors associated with a high lung shunt fraction include large tumor size, hepatic vein invasion, the presence of a transjugular intrahepatic portosystemic shunt (TIPS), and dysmorphic intratumoral vessels. In patients with tumors larger than 5 cm, the lung shunt fraction is likely to be low if there is no hepatic vein invasion, no TIPS, and no dysmorphic intratumoral vessels. Therefore, by selecting patients without dysmorphic intratumoral vessels for same-day TARE, it is possible to avoid wasting SIR-Spheres vials and perform the procedure without delays in treatment.

Furthermore, by defining safe and effective dose ranges for lung dose, tumor dose, and perfused liver dose, a standardized TARE protocol can be established. Through this study, we aim to establish appropriate patient selection criteria for same-day TARE and to standardize TARE dosimetry.

ELIGIBILITY:
Inclusion Criteria:

* HCC can be diagnosed by AASLD guideline
* hepatocellular carcinoma 5cm or larger
* dysmorphic intratumoral vessels 3mm or smaller
* Child-Pugh class A
* ECOG 0 or 1
* the following lab should be met. A. Leukocytes ≥ 1,000/µL and ≤ 20,000/µL B. Hemoglobin ≥ 6.0 g/dL (transfusion allowed to meet this criterion) C. Total bilirubin ≤ 2.0 mg/dL D. Platelet ≥ 40,000/µL E. International normalized ratio (INR) ≤ 2.0 for patients not taking anticoagulants F. Aspartate transaminase (AST) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) G. Alanine transaminase (ALT) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) H. Creatinine ≤ 2.5 mg/dL (if patient is receiving hemodialysis, no upper limit of creatinine)

Exclusion Criteria:

* hepatic vein invasion on CT/MRI
* hepatic vein enhancement on arterial phase of CT/MRI
* TIPS
* dysmorphic intratumoral vessels > 3mm
* main portal vein invasion
* significant COPD or interstitial lung disease
* biliary stent or enterobiliary anastomosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocellular carcinoma who are scheduled for radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of execution of same-day radioembolization procedure | Day 1
  Execution means that planning angiography, MAA scan and radioembolization are performed in a single day. The number same-day radioembolization is divided by total enrolled patient number.

SECONDARY OUTCOMES:
Objective response rate | up to 1 year
  objective response rate
local progression-free survival | From date of radioembolization until the date of first documented progression of treated tumor or date of death from any cause, whichever came first, assessed up to 60 months
Progression-free survival | From date of radioembolization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
overall survival | From date of radioembolization until the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi TW, Joo I, Kim HC. Association of dysmorphic intratumoral vessel with high lung shunt fraction in patients with hepatocellular carcinoma. Sci Rep. 2022 Aug 21;12(1):14248. doi: 10.1038/s41598-022-18697-5. PMID 35989374